CLINICAL TRIAL: NCT00003421
Title: A UKLG Randomised Trial of Initial Chemotherapy for Advanced Stage Hodgkins Disease
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066441; MRC-UKLG-LY09; EU-98020
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2007-05

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; ABVD protocol; Chlorambucil; Dacarbazine; Doxorubicin; Etoposide; Prednisolone; Procarbazine; Vinblastine; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: ABVD regimen
Drug: chlorambucil
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisolone
Drug: procarbazine hydrochloride
Drug: vinblastine sulfate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective for advanced Hodgkin's disease.

PURPOSE: Randomized phase III trial to compare different combination chemotherapy regimens in treating patients with advanced Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a four-drug anthracycline-based regimen or a seven-drug hybrid or eight-drug alternating regimen is the optimal treatment for patients with advanced Hodgkin's disease.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms. Arm I (ABVD): Patients receive doxorubicin IV, bleomycin IV, vinblastine IV, and dacarbazine IV on days 1 and 15. Courses repeat every 4 weeks. Arm II (ChlVPP/PABLOE): Patients receive oral chlorambucil, procarbazine, and prednisolone on days 1-14; vinblastine IV on days 1 and 8; doxorubicin IV on day 29; vincristine IV and bleomycin IV on days 29 and 36; oral etoposide on days 29-31; and oral prednisolone again on days 29-38. Courses repeat every 7 weeks. OR (Hybrid - ChlVPP/EVA): Patients receive vincristine IV on day 1; oral etoposide on days 1-5; oral chlorambucil, procarbazine, and prednisolone on days 1-7; and doxorubicin IV and vinblastine IV on day 8. Courses repeat every 4 weeks. Patients in both arms receive up to 6-8 courses of treatment. Radiotherapy may be given to sites of previous bulk disease for patients in complete remission or uncertain remission. Patients who achieve partial remission may receive radiotherapy to residual disease sites. Patients who fail to respond, or have disease progression, may receive induction therapy followed by high-dose consolidation therapy. Patients are followed every 3 months for 2 years, every 6 months for 5 years, and then annually for 5 years.

PROJECTED ACCRUAL: Approximately 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced Hodgkin's disease requiring systemic therapy Stage IA or IIA disease with bulky disease or more than three sites of involvement are also eligible

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other active malignancy within 5 years HIV negative Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for Hodgkin's disease Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for Hodgkin's disease Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1998-06; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry W. Hancock, MD, Study Chair — Cancer Research Centre at Weston Park Hospital
Locations (2):
- United Kingdom (2):
  - St. James's Hospital, Leeds, England
  - Weston Park Hospital, Sheffield, England

REFERENCES:
- [Result] Johnson PW, Radford JA, Cullen MH, Sydes MR, Walewski J, Jack AS, MacLennan KA, Stenning SP, Clawson S, Smith P, Ryder D, Hancock BW; United Kingdom Lymphoma Group LY09 Trial (ISRCTN97144519). Comparison of ABVD and alternating or hybrid multidrug regimens for the treatment of advanced Hodgkin's lymphoma: results of the United Kingdom Lymphoma Group LY09 Trial (ISRCTN97144519). J Clin Oncol. 2005 Dec 20;23(36):9208-18. doi: 10.1200/JCO.2005.03.2151. Epub 2005 Nov 28. PMID 16314615